CLINICAL TRIAL: NCT04536519
Title: Effects Of Foot Wear Modification Along With Physical Therapy On Functional Status In Knee Osteoarthritis
Brief Title: Foot Wear Modification Along With Physical Therapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Usman janjua, director Janjua rehab center, Isra University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1502-PHD-001
Record Dates: First submitted 2020-08-20; First posted 2020-09-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Osteo Arthritis Knee
Keywords: osteoarthritis; knee joint
MeSH Terms: conditions — Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial with 2 group
Who Masked: Participant, Care Provider
Masking Description: It was a double blinded study in which assessors and patientswere blinded. Close shoe type make it possible to blind patients because receiving identical conventional treatment in both groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Heel Wedged Insole Alone with physical therapy (Active Comparator): the lateral heel wedged insole (19) comprised non-custom, high density based on insoles of ethyl-vinyl acetate distributed bilaterally, preferably, covered in leather, were used in the study. The insole were equipped with a lateral wedge of 50 to 60.
  In the case of unilateral knee osteoarthritis, the non-wedge insole were used to compensate for possible leg length discrepancy in the contra-lateral leg. Shoes used was based on gymnast type to keep wedge insole in place. This further finalized individual to individual with unanimous decisions of Cordwainers, orthotics, and principal researcher, physiotherapist.
  Interventions: Other: osteoarthritis management
- Lateral aand medial Heel Wedged Insole with physiotherapy (Active Comparator): medial arch support part were combine with aforementioned lateral heel wedged support, full length support. There is a debate, however, 4 to 6 mm of full length support is considered to be effective for required alteration in mechanics
  Interventions: Other: osteoarthritis management

INTERVENTIONS:
Other: osteoarthritis management — The conventional physical therapy will be consisted of an array of protocols being deployed in parallel. This will consist of
  * Patient education regarding deforming forces, strategies of prevention and home exercise program
  * Decreasing stiffness by controlled active range of motion and mobilization techniques involving join play.
  * Mechanical stresses will be controlled in form of support provided by foot wear modification
  * Range of motion will be increased muscle stretches and manual mobilization techniques
  * Muscle performance and neuromuscular control will be addressed by gentle exercises of low intensity and repetitive exercises.
  * Balance improvement by employing balance training activities as part of treatment
  * Physical conditioning low impact or non-impact aerobics This conventional exercise will be given as baseline treatment to both of groups.
  Other Names: physical therapy

SUMMARY:
Orthotics and Prosthetics are important areas where physiotherapists order a variety of assistive aids to restore, compensate, or prevent physical ailments and disorders, such as here, Knee Osteoarthritis.

This study will be helpful not only in establishing the role of footwear modification as an adjunct treatment protocol for knee osteoarthritis but also elicit a multidisciplinary team approach which is a much-needed area, especially in the emergency rehabilitation area.

DETAILED DESCRIPTION:
2.1 MULTIDISCIPLINARY TEAM APPROACH As defined by World Health Organization, Curriculum Contents and International Practice Patterns, physical therapy is an autonomous profession where clinical make clinical decisions based on clinical reasoning, differentially diagnose, determine prognosis, and make plan of care including discharge planning and outcome assessment.

Orthotics and Prosthetics are important areas where physiotherapist order variety of assistive aids to restore, compensate or prevent physical ailments and disorders, such as here, Knee Osteoarthritis.

This study will be helpful not only establishing role of foot wear modification as adjunct treatment protocol for knee osteoarthritis but also elicit a multidisciplinary team approach which is a much needed area especially in emergency rehabilitation area.

2.2 LITERATURE GAP Although, there is work on performance of modified foot wears, which have been studied mostly alone or as adjunct with pharmacology. There is less literature on conservative treatment of osteoarthritis with foot wear modification coupled with physiotherapy treatment. This study will create a unique impact paying ways for type of preferable footwear that should be used, based on results, and combining treatment with physiotherapy care.

2.3 UNSETTLED DEBATE OVER TYPE OF FOOTWEAR The debate is still underway, worldwide, regarding which shoe type or foot wear should be preferred over other. The study results will come up with a contribution towards determining right foot wear for osteoarthritis.

2.4 COST EFFECTIVENESS The knee osteoarthritis is a problem that degenerative in nature and is triggered due to posture and abnormal force distribution. Right shoes are proven to alter walk posture, step length and degree of ease in walk. This simple remedy can be integral for reduction in care cost by minimizing disability and pain.

2.5 NOVEL SHOE MAKING APPROACH Although, advising foot wears and its modification is technical phenomenon, yet, this study can impact formulation of a shoe pattern that can help the arthritis patients. This can open new shoe making approach on public shoe outlets, from where old age individuals can directly buy the shoes that be the potential healer and disease modifier.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* diagnosed patient with knee osteoarthritis on clinical and radiographic basis,
* aged 50 years or above,
* knee pain from at least one month with an intensity equal or more than 4 on 11 points Numeric rating pain scale,
* falling between grade 2-3 on Kellgren-Lawrence Classification System for knee osteoarthritis,
* having BMI range between 22-25 kg/m2 and participating in study with their own will with a signed consent form.

Exclusion Criteria:

* trauma in knee region,
* having knee or lower limb surgery for fracture or arthroplasty,
* getting steroid based intra-articular injection or physiotherapy treatment in last 6 months,
* getting lidocaine intra-articular injection in last one month, with condition of systemic arthritic condition, severe co-morbidities or
* serious medical conditions or systemic disease causing dependent edema making difficult to wear foot wear in open or close shoes.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
knee osteoarthritis outcome score | 24 week
  questionaire used to evaluate charecteristics of knee joint
The Western Ontario and McMaster Universities Osteoarthritis Index | 24 week
  questionaire used to evaluate charecteristics of knee joint
Short Form 36 Health Survey Questionnaire | 24 week
  The Short Form 36 Health Survey Questionnaire (SF-36) is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions. Culture-specific data are required to calculate SF-36 norm-based scores.

SECONDARY OUTCOMES:
Manual Muscle Testing | 24 week
  muscle grading and power evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Janjua Rehab Center, Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Transcript and interview recording will be kept in a password protected environment. Identifying details will be taken out during data collection and analysis, any final report and any publication so people reading these will not able to identify these details. The documents pertaining to the administration of the research, such as consent form will be kept in a folder called project folder. This is a locked away security. People who are allowed to see the documents cannot pass this information to anyone else. All the documents will be destroyed after 7 years while audio recording will be erased after 2 years. Only staff involved in the data collection and analysis and people in authority will know the identity of the patients. Patients who will meet the criteria, their recruitment process will be kept secret only staff physiotherapist will know about it.